CLINICAL TRIAL: NCT03449329
Title: Randomised Controlled Double Blinded Trial Analyzing Impact of Serratus Intercostal Plane Block in Video Assisted Thoracic Surgery on Postoperative Pain and Recovery.
Brief Title: RCT Impact of Serratus Intercostal Plane Block in Video Assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, Head of department of anesthesiology,, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT impact of SIPblock
Record Dates: First submitted 2018-02-19; First posted 2018-02-28 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: double blinded randomized two study group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo SIP block (Placebo Comparator): This group will receive a placebo SIP block injection with 60mL NaCl 0.9%
  Interventions: Procedure: SIP
- Locoregional SIP block (Active Comparator): This group will receive a SIP block using:
  3mg/kg Ropivacain 1%
  1mcg/kg dexmedetomidine (Dexdor®) 100mcg/ml Addition of NaCl 0.9% up to 60ml
  Interventions: Procedure: SIP

INTERVENTIONS:
Procedure: SIP — The intervention group will receive a SIP block

SUMMARY:
Rationale Video Assisted Thoracic Surgery (VATS) is known to be a moderate painful procedure. There are many ways to manage postoperative pain following this kind of surgery. One of the 'golden standards' nowadays is epidural analgesia using Patient Controlled Epidural Analgesia (PCEA). Patient Controlled Intravenous Analgesia (PCIA) is also an option, as are several kinds of regional anesthesia. One of the most recent described regional blocks is the Serratus Anterior Plane block (SAP), also called Serratus Intercostal Plane (SIP) block.

Objectives The objective of this study is to evaluate the efficacy and opioid sparing effect of a SIP block in postoperative pain relief after VATS.

Hypotheses Patients receiving a SIP block prior to surgery need less opioids during and 24h after VATS compared with patients who didn't receive a SIP block.

Study design Single center randomized controlled trial Study population Patients older than 18 years old scheduled for VATS. Main study parameters/endpoints The primary endpoint is the opioid use during the first 24 hours after start of surgery. Secondary endpoints are the VAS score on day 0 and day 1 after surgery, and the prevalence of postoperative nausea and vomiting (PONV).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness In the intra-operative period, patients will not experience discomfort from either strategy because of general anesthesia. If the hypothesis proves to be true, patients with SIP block could benefit from a lower amount of received opioids, which could give less chance of opioid associated adverse effects. There won't be any additional blood sampling related to this study.

DETAILED DESCRIPTION:
The proposed randomized controlled trial aims at comparing the opioid use per- and postoperatively in patients with versus without SIP block undergoing VATS.

We hypothesize that use of a SIP block results in less opioid use during and the first 24 hours after VATS as compared with patients without SIP block.

Single center randomized controlled trial on patients undergoing VATS under general anesthesia.

We intend to recruit patients scheduled for elective VATS in our hospital during a period of 3 months. Surgical patients will be screened twice a week, because there are two days a week that VATS procedures take place in our hospital. We will randomize 20 patients, based on the power analysis (cfr infra).

Inclusion criteria: Patients scheduled for VATS under general anesthesia Exclusion criteria

* Age < 18 years
* Urgent surgery
* Allergy to sufentanil or ropivacain
* Postoperative need for invasive ventilation within 24hours after surgery

Sample size calculation was based on our primary hypothesis and primary study outcome, and was informed by data collected in patients who underwent VATS procedures in our hospital during the previous six months. These calculations indicate that 14 patients need to be included, assuming a significance level of 0.05 and a power of 80%, to detect the expected difference in per- and postoperative opioid use between the SIP-group and the placebo group.

Main study parameter/endpoint: Opioid use during the first 24 hours after end of surgery Secondary study parameters/endpoints

* VAS score on day 0 and day 1
* Postoperative nausea and vomiting (PONV)

Surgical patients in our hospital will be considered eligible if they fulfill the entry criteria. Eligible patients will be screened, their demographic data recorded (registry: age, gender, type of surgery) and those without exclusion criteria will be randomized. In total, 20 patients will be included.

Patient Consent All patients or legal guardians must provide written informed consent according to local regulations before inclusion in the study.

Randomization will be performed using a sealed envelope system. Randomization arms Before surgery patients will be randomly assigned 1:1 to a placebo SIP block or to a real SIP block. All investigators involved intra- and postoperative are blinded. An independent anesthesia nurse not involved peri-operatively is asked to prepare the drugs in a different location according to the info kept in a sealed envelope. This envelope remains sealed in the patient files to be broken if an adverse event happens.

After induction of anesthesia and before surgery, each patient will receive an injection in between the serratus anterior and the intercostal muscle. The injection will be localized in the midaxillary line, between the 4th and 5th rib. The intervention group will receive a total amount of 60cc which consists of:

* 3mg/kg Ropivacain 1%
* 1mcg/kg dexmedetomidine (Dexdor®) (ampul with 2 ml contains 100mcg/ml)
* Addition of NaCl 0.9% up to 60ml The control group will receive an injection of 60cc NaCl 0.9% at the same injection site of the SIP block.

Each patient will receive 5-15mcg sufentanil (Sufenta®) before induction of anesthesia, depending on the personal choice of the anesthesiologist. To induce anesthesia, patients will receive 2mg/kg propofol 1% (Propofol®), and if not sufficient, a supplemental bolus will be given. To receive adequate neuromuscular blockage, at least 0.6mg/kg rocuroniumbromide 1% (Esmeron®) will be used.

Starting from insicion, depending on the personal choice of the performing anesthesiologist or based on ANI monitoring, a supplemental bolus sufentanil will be given if considered necessary. Routine intra-operative monitoring should include noninvasive blood pressure measurements, pulse oximetry, end-tidal carbon dioxide fraction and electrocardiography. Every patient should receive at least one peripheral venous line to allow adequate fluid resuscitation during the study period. Nasogastric tubes, urinary bladder catheters and/or other intravenous catheters, as well as other, more invasive monitoring may be used according to local practice and/or guidelines.

All patients receive a PCIA pump with sufentanyl and the dose requested and given is measured for the first and the second day. Patients receive paracetamol 1 gram every 6 hours.

Data to be collected

Pre-operative variables will be collected at the pre-anesthetic visit or before induction of general anesthesia:

Intra-operative variables will be collected after induction of anesthesia and during surgery:

Postoperative variables will be collected with a patient questionnaire and clinical examination, both on day 0 en 1 after surgery. Following variables will be collected:

Patient characteristics will be compared and described by appropriate statistics. The analysis will be performed with STATA or SPSS.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for thoracoscopic surgery

Exclusion Criteria:

* urgent surgery
* allergic to Sufentanil or Ropivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Opioid consumption during the first 24 hours postoperative | first 24 hours postoperative (after wound closure)
  total dose of opioids given

SECONDARY OUTCOMES:
Intraoperative opioid consumption | intra operative (from incision till wound closure)
  total dose of opioids used intra operative

CONTACTS AND LOCATIONS:
Overall Officials: Marco Lanckneus, MD, Study Chair — AZ Sint Jan Brugge-Oostende
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No